CLINICAL TRIAL: NCT04461977
Title: Acupuncture for Treatment of Peripheral Neuropathy Induced by Neoadjuvant or Adjuvant Paclitaxel in Early Stage Breast Cancer: a Sham Controlled, Randomized Study
Brief Title: Acupuncture for Peripheral Neuropathy Induced by Paclitaxel in Early Stage Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Brasileiro de Controle do Cancer (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 26778919.3.0000.0072
Record Dates: First submitted 2020-07-02; First posted 2020-07-08 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Peripheral Neuropathy Due to Chemotherapy
Keywords: Peripheral Neuropathy; Breast Cancer; Chemotherapy; Paclitaxel; Acupuncture
MeSH Terms: conditions — Peripheral Nervous System Diseases; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: True acupuncture vs sham acupuncture
Who Masked: Participant
Masking Description: Sham acupuncture
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A - true acupuncture (Experimental): The selection of acupuncture points is based on Traditional Chinese Medicine (Wen 2011) and on previous studies (Jeong, 2018; Bao,2018), selected as main points: bilateral "baxie", SJ5, "bafeng", KID3 and ST36. Modifications or additional secondary points may be indicated according to clinical judgment throughout treatment.
  Interventions: Other: True acupuncture
- B - sham acupuncture (Sham Comparator): Patients will receive needling at non-acupuncture points with superficial needling without manipulation to obtain "de qi", located near the real points in the hands and feet.
  Interventions: Other: Sham acupuncture

INTERVENTIONS:
Other: True acupuncture — The selection of acupuncture points is based on Traditional Chinese Medicine (Wen, 2011) and on previous studies (Jeong,2018; Bao,2018), selected as main points: bilateral "baxie", SJ5, "bafeng", KID3 and ST36. Modifications or additional secondary points may be indicated according to clinical judgment throughout treatment. The needles will be inserted at a depth of 10 - 15 mm, being gently manipulated to obtain "de qi" sensation. The needles will be left for 20 - 25 minutes. There will be once a week acupuncture treatment, for 8 consecutive weeks. The acupuncture needles will be sterile, disposable stainless steel needles size 0.20 x 30 mm, of Korean brand Dong Bang, Chungcheongnam-do.
  Arms: A - true acupuncture
Other: Sham acupuncture — Patients will receive needling at non-acupuncture points with superficial needling without manipulation to obtain "de qi", located near the real points in the hands and feet. The needles will also be left for 20 - 25 minutes. There will be once a week acupuncture treatment, for 8 consecutive weeks. There will be once a week acupuncture treatment, for 8 consecutive weeks. The acupuncture needles will be sterile, disposable stainless steel needles size 0.20 x 30 mm, of Korean brand Dong Bang, Chungcheongnam-do.
  Arms: B - sham acupuncture

SUMMARY:
The present study aims to evaluate the effectiveness of acupuncture in the treatment of chemotherapy drug paclitaxel induced peripheral neuropathy in patients with early stage breast cancer

DETAILED DESCRIPTION:
Patients with early stage breast cancer (stages I,II,III) who received paclitaxel in neoadjuvant or adjuvant chemotherapy protocol and developed peripheral neuropathy will be randomized to receive true acupuncture (intervention group) vs sham acupuncture (control), once a week, for 8 weeks. The primary outcome is improvement of the symptoms by Neuropathic Pain Symptom Inventory (NPSI) scale (Bouhassira,2004). The secondary outcomes are improvements on Visual analog scale (VAS) and Quality of life by FACT-taxane (Cella, 2003) questionnaire. These scales will be assessed in the Screening visit (baseline), week 4, week 6, week 8 and week 12. The study has duration of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old.
* Agreed to sign the Informed Consent Term
* ECOG 0-1
* Breast cancer stages I, II and III.
* Received adjuvant or neoadjuvant chemotherapy containing weekly paclitaxel 80 mg/m2.
* Peripheral sensory neuropathy grade 2 and 3 by the "Common Terminology Criteria for Adverse Events" (CTCAE) v5.0

Exclusion Criteria:

* Previous history of peripheral neuropathy due to other comorbidities.
* Prior treatment with chemotherapy for cancer other than breast cancer.
* Use of medications to treat peripheral neuropathy.
* Metastatic disease.
* Presence of lymphedema of any degree.
* History of coagulopathy or full anticoagulation.
* Previous acupuncture treatment for any indication within the last 90 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
The change the effects of neuropathic pain syndromes management from baseline | Screening visit (baseline), week 4, week 6, week 8, week 12
  Neuropathic Pain Symptom Inventory (NPSI) scale. This tool included 12 items in total: 10 are differential symptoms descriptors and 2 items evaluate spontaneous and paroxysmal spontaneous pain. The verbal numeric scale from zero (no pain) to 10 (worst imaginable pain). Total pain intensity score may be calculated by the sum of 10 descriptors.

SECONDARY OUTCOMES:
Baseline pain intensity change | Screening visit (baseline), week 4, week 6, week 8, week 12
  Visual analog scale (VAS). The pain VAS is a unidimensional measure of pain intensity. It is a continuous scale comprised of a horizontal (HVAS) or vertical (VVAS) line, usually 10 centimeters (100 mm) in length. For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]).
Change in side effects associated with taxane treatments from baseline | Screening visit (baseline), week 4, week 6, week 8, week 12
  FACT-taxane questionnaire. It is a self-report instrument that was developed to measure the health-related Quality of life of patients receiving taxane-containing chemotherapy. This scale has 16 items, including an 11-item neurotoxicity subscale and five additional taxane-specific questions related to the effects of arthralgia, myalgia, and skin changes. The total score is calculated as the sum of the un-weighted subscale score.

CONTACTS AND LOCATIONS:
Overall Officials: Lin I Ter, MD, Principal Investigator — Instituto Brasileiro de Controle do Cancer
Locations (1):
- Instituto Brasileiro de Controle de Cancer (IBCC Oncologia), São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bouhassira D, Attal N, Fermanian J, Alchaar H, Gautron M, Masquelier E, Rostaing S, Lanteri-Minet M, Collin E, Grisart J, Boureau F. Development and validation of the Neuropathic Pain Symptom Inventory. Pain. 2004 Apr;108(3):248-257. doi: 10.1016/j.pain.2003.12.024. PMID 15030944
- [Background] Cella D, Peterman A, Hudgens S, Webster K, Socinski MA. Measuring the side effects of taxane therapy in oncology: the functional assesment of cancer therapy-taxane (FACT-taxane). Cancer. 2003 Aug 15;98(4):822-31. doi: 10.1002/cncr.11578. PMID 12910528
- [Background] Jeong YJ, Kwak MA, Seo JC, Park SH, Bong JG, Shin IH, Park SH. Acupuncture for the Treatment of Taxane-Induced Peripheral Neuropathy in Breast Cancer Patients: A Pilot Trial. Evid Based Complement Alternat Med. 2018 Oct 21;2018:5367014. doi: 10.1155/2018/5367014. eCollection 2018. PMID 30420895
- [Background] Bao T, Seidman AD, Piulson L, Vertosick E, Chen X, Vickers AJ, Blinder VS, Zhi WI, Li Q, Vahdat LT, Dickler MN, Robson ME, Mao JJ. A phase IIA trial of acupuncture to reduce chemotherapy-induced peripheral neuropathy severity during neoadjuvant or adjuvant weekly paclitaxel chemotherapy in breast cancer patients. Eur J Cancer. 2018 Sep;101:12-19. doi: 10.1016/j.ejca.2018.06.008. Epub 2018 Jul 13. PMID 30007894
- [Background] de Andrade DC, Ferreira KA, Nishimura CM, Yeng LT, Batista AF, de Sa K, Araujo J, Stump PR, Kaziyama HH, Galhardoni R, Fonoff ET, Ballester G, Zakka T, Bouhassira D, Teixeira MJ. Psychometric validation of the Portuguese version of the Neuropathic Pain Symptoms Inventory. Health Qual Life Outcomes. 2011 Nov 30;9:107. doi: 10.1186/1477-7525-9-107. PMID 22128801
- [Background] Wen TS. Acupuntura Clássica Chinesa. Edição Dig. São Paulo: Cultrix; 2011.
- [Derived] Ter LI, Yamada AMTD, do Nascimento Martins Basilio A, Lopez RVM, Hsing WT. Acupuncture for peripheral neuropathy induced by paclitaxel in early-stage breast cancer: a randomized, parallel, controlled, blinded study in a Brazilian Oncologic Center (PACLILIN Study). Support Care Cancer. 2026 Jan 16;34(2):102. doi: 10.1007/s00520-026-10315-8. PMID 41543601
- See also: Common Terminology Criteria for Adverse Events ( CTCAE ) version 5.0. — https://ctep.cancer.gov/protocolDevelopment/electronic_applications/docs/CTCAE_v5_Quick_Reference_8.5x11.pdf